CLINICAL TRIAL: NCT04034537
Title: Repository of Phase Signals for Algorithm Development and Testing in Subjects With Coronary Artery Disease in China
Brief Title: Repository of Phase Signals for Algorithm Development and Testing in CAD in CHINA
Acronym: CADChina
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CADC-CIP-001
Record Dates: First submitted 2019-07-21; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; cardiac Phase Space Tomography Analysis; ischemia
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Intervention Model Description: All patients are planned to perform coronary angiography without contraindications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cPSTA GROUP (Experimental): Patients who meet the study's inclusion and exclusion criteria, including signing the informed consent form, subjects will undergo cardiac Phase Space Tomography Analysis (cPSTA) signal acquisition prior to their scheduled cardiac catheterization on the day of the procedure.
  Interventions: Diagnostic Test: cPSTA

INTERVENTIONS:
Diagnostic Test: cPSTA — The cPSTA System is a medical device system that uses passive tomography to analyze a patient's phase space data to identify the presence of significant coronary artery disease. The cPSTA System consists of several components that work together to obtain, transmit, analyze the data, and display the results, including the Phase Signal Acquisition System (PSAQ System), which is the Phase Signal Recorder (PSR) and the Phase Signal Data Repository (PSDR); analytical software; and secure web portal. For this study only the PSAQ System is used by the clinical site for the purposes of acquiring and transmitting the signal. All enrolled patients will perform cPSTA signal recording.
  Other Names: PSR

SUMMARY:
The primary objective of this study is to build a repository of resting cardiac phase space signals from eligible subjects using the Phase Signal Recorder (PSR) prior to coronary angiography for the purposes of machine-learning and testing algorithms developed by Analytics 4 Life. Male and Female subjects will be uniquely and consecutively enrolled into one group to support populating a repository of phase signals.

DETAILED DESCRIPTION:
Analytics 4 Life (A4L) is a medical information technology company that uses advanced signal processing techniques for the purposes of assessing and diagnosing disease. A4L is currently focused on developing a non-invasive solution for the assessment of significant coronary artery disease using the cardiac Phase Space Tomography Analysis (cPSTA) System. Through proprietary variable extraction to define phase space signals as metrics in mathematical terms and machine learned formulas, A4L has developed a cost-effective solution to collect and analyze phase signals as data indicative of cardiac performance. The cPSTA System passively reconstructs and displays images from this data using topological data analysis (TDA) to provide a computationally tractable method of interrogating the complex physiological processes of the heart with the intent to understand and characterize the cardiac tissue properties.

A4L has providing the Phase Signal Recorder (PSR) to the sponsor for use in this study. The primary objective of this study is to collect resting phase signals from eligible subjects using the Phase Space Recorder (PSR) prior to coronary angiography for the purpose of machine learning and testing an algorithm developed to assess the presence of significant coronary artery disease (CAD).The definition of significant CAD, which is well established in the literature, is either the presence of a stenosis ≥50% by angiography or reduced blood flow of <0.80as measured by Fractional Flow Rate (FFR) or instantaneous free-wave ratio (iFR) <0.89.Each subject's CAD status will be assessing the presence of significant CAD in the major coronary arteries including the left main artery (LMA), left anterior descending artery (LAD), circumflex artery (LCX), and the right coronary artery (RCA) and their distributions.

Accurately assessing the presence or absence of CAD and evaluating other physiologic measures is vital to the assessment of cardiac health/illness. As such, the following additional assessments are planned to support further support goal: establishing a ROC curve for the primary objective to describe a full range of sensitivity and specificity trade-offs; and, developing and testing machine-learned algorithms to validate a clinically relevant sensitivity and specificity for the identification of significant CAD specific to perfusion regions (LAD, LCX, and RCA).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old
2. Meets criteria for coronary angiography
3. Scheduled to undergo cardiac catheterization with coronary angiography
4. Ability to understand the requirements of the study and to provide written informed consent

Exclusion Criteria:

1. Prior coronary artery bypass grafting (CABG)
2. Prior heart valve replacement
3. Previous sustained or paroxysmal atrial or ventricular arrythmia;
4. Infiltrative myocardial disease (amyloid, sarcoid, right ventricular dysplasia);
5. Presence of cardiac implantable electronic device (CIED), including implantable cardioverter defibrillator (ICD), pacemaker (PM), implantable loop recorders and other monitors
6. Implantable Neuro-stimulators
7. Congenital Heart Disease
8. Pregnant or breast feeding
9. Currently taking any Type IA, IC or III antiarrhythmics
10. Any history of amiodarone use
11. Clinically significant chest deformity (e.g., pectus excavatum or pectus carinatum)
12. Breast implants
13. Neuromuscular Disease if the condition results in tremor or muscle fasciculations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
positive coronary artery disease | 7 day after index procedure
  significant stenosis measured by coronary angiography
positive cardiac Phase Space Tomography Analysis | 7 day after index procedure
  positive result measured by cardiac Phase Space Tomography Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Juying Qian, M.D., Principal Investigator — Shanghai Zhongshan Hospital

IPD SHARING:
Plan to Share IPD: No